CLINICAL TRIAL: NCT02694211
Title: Stress Prevention at Work: Intervention Efficacy and Implementation Process Evaluation (SPA)
Brief Title: Stress Prevention at Work: Intervention Efficacy and Implementation Process Evaluation
Acronym: SPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Irene Jensen, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2012/2200-31/5
Record Dates: First submitted 2014-09-30; First posted 2016-02-29 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Stress, Psychological
Keywords: work related stress
MeSH Terms: conditions — Stress, Psychological; Occupational Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group ProMES (Experimental): Productivity measurement and enhancement system (ProMES) is a participatory intervention for productivity enhancement. Core strategies of this method could be addressing known work stressors such as absence of influence and control, insufficient interaction with coworkers, unclear and conflicting tasks, insufficient participation in decision-making and insufficient feedback
  Interventions: Behavioral: ProMES
- Control group (No Intervention): No intervention, business as usual

INTERVENTIONS:
Behavioral: ProMES — Productivity measurement and enhancement system (ProMES) is a participatory intervention for productivity enhancement. Core strategies of this method could be addressing known work stressors such as absence of influence and control, insufficient interaction with coworkers, unclear and conflicting tasks, insufficient participation in decision-making and insufficient feedback
  Arms: Intervention group ProMES

SUMMARY:
The Stress prevention at work (SPA) project intends to evaluate the method named Productivity Measurement and Enhancement System (ProMES) as a stress preventive approach among health care employees.

DETAILED DESCRIPTION:
Stress-related illnesses are today together with musculoskeletal disorders the predominant cause of production loss and absenteeism. The risks of developing stress-related mental illness is today well established, however, it is less studied how this can be successfully treated or prevented in workplaces through interventions.

The SPA project intends to evaluate the method the Productivity Measurement and Enhancement System (ProMES). The method is mainly evaluated for production improvement, but there are indications that it also has stress-reducing effect on working groups. The method gives employees within health care opportunities to participate actively in productivity-enhancing measures. The employees, along with their immediate supervisors, identify and prioritize responsive and desirable results in all of the activities important dimensions. International studies have shown that participation (participation) has positive effects on employee performance and attitudes.

The aim of this study is to test whether efforts in targeting the organization and work environment can reduce stress and prevent stress-related ill health in the workplace. Primary outcomes of the study are tense work i.e. imbalance between demand and control and other primary indicators of stress, such as sleep and recovery.

The hypothesis in study 1 is that productivity enhancing workplace interventions based on a participative approach also increases employees' sense of control and control over their own work. This in turn means that the method also could be used to reduce the occurrence of tense work and thus affect / reduce the stress-related illness.

ELIGIBILITY:
Inclusion Criteria:

* All employees (18-67 years) employed at the intervention and control primary care units, who were actually working at the time for this study

Exclusion Criteria:

* employees absent due to long-term illness,
* employees absent due to parental leave
* employees absent due to long-term studies

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2013-05; Primary Completion 2014-10 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change in job strain (a measure of the balance between job demand and job control) | baseline, 6-months, 12-months
  QPSNordic questionnaire

SECONDARY OUTCOMES:
Change in Effort-Reward Imbalance | baseline, 6-months, 12-months
  Effort-Reward Imbalance Questionnaire
Change in experience of stress | baseline, 6-months, 12-months
  Single item stress question from Elo, A-L., Leppänen, A., Lindström K., Ropponen, T. OSQ-Occupational Stress Questionnaire: user's instructions. Helsinki: Finnish Institute of Occupational health; 1992. Reviews 19.
change in sleep difficulties | baseline, 6-months, 12-months
  Two single questions Reference: Åkerstedt, T., Knutsson, A., et al. 2002. Att predicera sömnstörning, insomningsrisk och mental trötthet - tre delstudier. Psykosocial belastning och riskfaktorer för hjärtkärlsjukdom. Arbete och Hälsa 2002:7. Westerholm, P. Stockholm, Arbetslivsinstitutet
change in Recovery | baseline, 6-months, 12-months
  One single question. Reference: Aronsson, G. och Svensson, L. 1997. Nedvarvning, återhämtning och hälsa bland lärare i grund- och gymnasieskolan. Arbete och Hälsa 1997:21. Stockholm, Arbetslivsinstitutet.
change in depression | baseline, 6-months, 12-months
  Hospital Anxiety and Depression Scale
change in Sick leave | baseline, 6-months, 12-months
  One single question:How many working days during the last 7 days, have you been away from work because of sick leave?
change in General health | baseline, 6-months, 12-months
  A question from General Health Questionnaire (WHO)
change in Productivity | baseline, 6-months, 12-months
  Questions from "Measuring production loss due to health and work environment problems: construct validity and implications."(Report) Lohela Karlsson, Malin ; Hagberg, Jan ; Bjorklund, Christina ; Bergstrom, Gunnar ; Jensen, Irene Journal of Occupational and Environmental Medicine, Dec, 2013, Vol.55(12), p.1475(9). Karolinska institutet. Stockholm
change in Exhaustion | baseline, 6-months, 12-months
  Oldenburg Burnout Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Irene Jensen, Professor, Principal Investigator — Karolinska Institutet

IPD SHARING:
Plan to Share IPD: No